CLINICAL TRIAL: NCT04283877
Title: The Role of Methylphenidate on Performance in the Cold
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Brock University (Other)
Responsible Party: Principal Investigator, Stephen Cheung, Professor, Brock University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: EEL124
Record Dates: First submitted 2019-09-13; First posted 2020-02-25 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Hypothermia; Exercise Test; Cognition
MeSH Terms: conditions — Hypothermia | interventions — Methylphenidate

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Who Masked: Investigator
Masking Description: Double-blinding of participants and investigator, with independent investigator in charge of placebo and drug
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Methylphenidate (Experimental): 30 mg methylphenidate, 60 minutes before testing
  Interventions: Drug: Methylphenidate
- Control (Placebo Comparator): 30 mg of lactose pill, 60 minutes before testing
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Methylphenidate — 3 x 10 mg oral tablets. Single acute dose for all participants
  Arms: Methylphenidate
Drug: Placebo oral tablet — 3 x 10 mg oral lactose tablet for all participants
  Arms: Control

SUMMARY:
The purpose is to study the effects of dopamine activity, using methylphenidate ingestion, on exercise and cognitive function over the course of a progressive cooling protocol. The investigators hypothesize that methylphenidate will minimize the previously reported impairment in exercise performance and cognitive function with mild hypothermia and cold stress (air temperature: 0˚C) compared to placebo, suggesting that dopamine activity preserves exercise and cognitive capacity with mild hypothermia.

DETAILED DESCRIPTION:
Temperature regulation and decision-making are vital aspects of human survival where relatively small deviations in whole-body heat balance lead to decrements in physical performance and cognitive function. Prolonged exposure to cold stress combined with inadequate clothing and/or insufficient heat production can lead to decreases in body temperature causing mild hypothermia (≤ -1.0˚C in body temperature). Performance in the cold is more physically demanding compared to neutral environments (~22˚C) as there is increased cardiovascular strain due to a strong peripheral vasoconstriction reducing cerebral and muscle blood flow and oxygenation, reduced neuromuscular capacity, as well as changes in energy metabolism during shivering and increased catecholamine release. Additionally, there is an increased psychological strain where perceptually there is a high thermal discomfort, alterations in neurotransmitters (e.g. dopamine, norepinephrine), and alterations in mood. These changes lead to decreases in self-paced cycling time-trial performance in the cold with mild hypothermia compared to thermoneutral environments. Additionally, there appears to be task-dependent cognitive changes with acute cold stress, where higher-order functions such as executive function, working memory, and inhibitory control decrease before simple task performance such as reaction time and visual recognition/awareness. Currently, it is unknown what the potential mechanisms are that lead to these performance decrements.

The decrements in both self-paced exercise and cognitive function may be due to alterations in neurotransmitters caused by hypothermia. Exposure to cold leads to alterations in dopamine, and norepinephrine which may affect prefrontal cortex function, which may explain why higher-order executive function tasks such as inhibitory control and spatial planning are impaired compared to simple task performance. Previously, it has been determined that the use of tyrosine (amino acid precursor to dopamine and norepinephrine neurotransmitters) supplementation improves working memory and executive function despite a -2.0˚C drop in body temperature through cold-water immersion, but not in thermoneutral conditions. However, it is unknown what the role of dopamine or central nervous system stimulants are in the cold. Methylphenidate is a central nervous system stimulant through dopamine re-uptake inhibition is demonstrated to improve executive function task performance in healthy adults in thermoneutral conditions. Additionally, methylphenidate has been demonstrated to improve self-paced cycling performance by 16% in the heat (30˚C) but not thermoneutral environments (1). Methylphenidate is also demonstrated to improve maximal force production during fatiguing exercise, indicating it may play a role in reducing the effects of fatigue during endurance exercise. The investigators aim to determine the role of the central nervous system using methylphenidate on cognitive function and self-paced exercise in the cold.

ELIGIBILITY:
Inclusion Criteria:

* Males and females

Exclusion Criteria:

* Diagnosed cardiovascular, respiratory, and/ or neuromuscular disease
* Prescription of MPH or any drugs for hyperactivity within the past 1 year
* Diagnosed mental health condition (e.g. depression, anxiety disorder)
* Raynaud's Disease or Cold Urticaria
* Current prescription medication (except for asthma or allergy medication)
* Pregnancy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-12-15 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
20 km cycling time trial | 2-4 hours post ingestion
  completion time in minutes
Cognitive function | 1-4 hours after ingestion
  mean reaction time in ms
cognitive function | 1-4 hours post ingestion
  # of errors made

CONTACTS AND LOCATIONS:
Locations (1):
- Environmental Ergonomic Laboratory - Brock University, St. Catharines, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
We will not be sharing individual participant data with other researchers.